CLINICAL TRIAL: NCT00107159
Title: A Phase II Study Of Matured Dendritic Cells Pulsed Ex Vivo With 3 Melanoma Cell Line Lysates (IDD-3) in Patients With In-Transit or Metastatic Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Unresected Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000422429; UCLA-0408080-01; IDM-DC-MEL-202
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-04

CONDITIONS: Melanoma (Skin)
Keywords: recurrent melanoma; stage III melanoma; stage IV melanoma
MeSH Terms: conditions — Melanoma

INTERVENTIONS:
Biological: autologous dendritic cell-allogeneic melanoma tumor cell lysate vaccine

SUMMARY:
RATIONALE: Vaccines made from a person's white blood cells and a donor's tumor cells may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase II trial is studying how well vaccine therapy works in treating patients with unresected stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the clinical activity of vaccine therapy comprising autologous dendritic cells pulsed with allogeneic melanoma tumor cell lysates (IDD-3), as measured by tumor control, in patients with unresected stage IIIB or IIIC or stage IV melanoma.

Secondary

* Determine the immunologic activity of this vaccine, as measured by T-cell and antibody responses to lysate or to melanoma antigens or peptides, in these patients.
* Determine the safety of this vaccine, as measured by the incidence and severity of adverse events, in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients undergo apheresis to collect peripheral blood mononuclear cells (PBMCs). The PBMCs are cultured with sargramostim (GM-CSF) and interleukin-13 for the production of dendritic cells. The dendritic cells are then pulsed with lysates from 3 allogeneic melanoma tumor cell lines (IDD-3) to produce the vaccine.

Patients receive vaccine therapy comprising IDD-3 administered as 1 subcutaneous and 5 intradermal injections at each of the 2 uninvolved lymph node-bearing regions once in weeks 0, 2, 4, 6, 8, 10, 16, and 22 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 2, 10, 18, and 26 weeks.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study within 4-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary cutaneous or unknown primary melanoma, including 1 of the following stages:

  * Stage IIIB or IIIC disease

    * Unresected, in-transit lymph node metastases (N2c or N3)
  * Stage IV disease

    * Distant skin, subcutaneous, lymph node, or pulmonary metastases (M1a or M1b)

      * No cerebral, bone, or other visceral metastases
* At least 1 measurable or evaluable lesion

  * Small-volume multiple cutaneous deposits allowed
* Progressive disease, as defined by 1 of the following criteria:

  * At least 20% increase in size in ≥ 1 measurable or evaluable lesion
  * Appearance of ≥ 1 new lesion since or during last treatment (if applicable) AND within the past 3 months

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 6 months

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10.0 g/dL (transfusion allowed)

Hepatic

* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN)
* Lactic dehydrogenase normal
* No active hepatitis B or C infection

Renal

* Creatinine ≤ 1.5 times ULN

Immunologic

* No history of autoimmune disease

  * Vitiligo allowed
* No history of immunodeficiency syndrome
* No active bacterial, viral, or fungal infection within the past 72 hours
* HIV-1 or -2 negative
* Human T-cell lymphotrophic virus-I or -II negative

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No contraindication to apheresis
* No other significant medical or surgical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior vaccine therapy with ≥ 1 melanoma antigen or peptide
* More than 4 weeks since prior biologic therapy

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy

* No concurrent chronic systemic corticosteroids

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* More than 4 weeks since prior investigational products
* More than 4 weeks since prior chronic systemic immunosuppressive treatment
* No concurrent medication or treatment regimen that would prelude study participation
* No other concurrent anticancer treatment
* No other concurrent immunosuppressive treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2005-01; Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Tumor control rate (complete response, partial response, or stable disease) for 4-8 weeks

SECONDARY OUTCOMES:
Safety
Immune response

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Ribas, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] Ribas A, Camacho LH, Lee SM, Hersh EM, Brown CK, Richards JM, Rodriguez MJ, Prieto VG, Glaspy JA, Oseguera DK, Hernandez J, Villanueva A, Chmielowski B, Mitsky P, Bercovici N, Wasserman E, Landais D, Ross MI. Multicenter phase II study of matured dendritic cells pulsed with melanoma cell line lysates in patients with advanced melanoma. J Transl Med. 2010 Sep 27;8:89. doi: 10.1186/1479-5876-8-89. PMID 20875102